CLINICAL TRIAL: NCT00551538
Title: Twenty-Four-Hour Plasma Glucose Profiles Observed in Patients With Type 2 Diabetes During Therapy Consisting of Oral Agent(s) Plus Twice-Daily Insulin Lispro Low Mixture or Once-Daily Insulin Glargine
Brief Title: 24 Hour Plasma Glucose Profiles Comparing Lispro Mix 75/25 vs. Glargine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7505; F3Z-MC-IOOM
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Diabetic; Insulin; Glargine; Lispro
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lispro mixture 75/25 twice-daily, SC injection, given in conjunction with oral antidiabetic medications.
  Interventions: Drug: Lispro mix 75/25
- 2 (Active Comparator): Glargine, once-daily, SC injection, given in conjunction with oral antidiabetic medications.
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Lispro mix 75/25 — Lispro mix 75/25 twice-daily, SC injection, given in conjunction with oral antidiabetic medications.
  Arms: 1
Drug: Glargine — SC injection, once-daily, given in conjunction with oral antidiabetic medications.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if twice-daily Lispro low mixture (75/25) will result in lower post prandial blood glucose readings versus once-daily glargine plus oral diabetic medications.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that a twice daily insulin regimen consisting of insulin lispro (mix 75/25)plus OAMs will result in a lower 2 hour postprandial plasma glucose, averaged across the morning and evening meals, compared with once daily insulin glargine plus OAMs at bedtime following 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have inadequate overall glycemic control (hemoglobin A1c greater than or equal to 7.0% and less than or equal to 12.0%) at or within 4 weeks prior to Visit 1
* Have used:

  * single or multiple OAMs for at least 3 months immediately prior to entering the study, including metformin, sulfonylurea, meglitinides (repaglinide, nateglinide), or alpha glucosidase inhibitors (acarbose, miglitol); or
  * insulin (once or twice daily) for at least 3 months immediately prior to entering the study; or
  * a combination of the above.
* Are greater than or equal to 21 and less than 80 years of age
* As determined by the investigator, are capable and willing to:

  * comply with their prescribed diet and medication regimen,
  * perform self blood glucose monitoring,
  * use the patient diary as required for this protocol,
  * participate in two 24 hour inpatient assessments

Exclusion Criteria:

* Have used a thiazolidinedione (pioglitazone or rosiglitazone) during the 3 months prior to entry into the study
* Are currently treated with a meglitinide without sulfonylurea
* Have a known allergy or intolerance to insulin lispro mix 75/25, insulin glargine, or metformin
* Have plasma creatinine greater than or equal to 1.5 mg/dL (for males) or greater than or equal to 1.4 mg/dL (for females) for patients who will be treated with metformin or; greater than 2 mg/dL for patients treated with other OAMs, as determined by a local laboratory
* Have received chronic (lasting longer than 2 weeks), systemic glucocorticoid therapy (excluding topical and inhaled preparations) within 4 weeks immediately prior to Visit 1

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-05; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Combined morning and evening mean 2 hour postprandial plasma glucose during each 24 hour inpatient period. | At end of treatment arm or 3 months.

SECONDARY OUTCOMES:
HbA1c | At end of treatment arm or 3 months.
2 hour plasma glucose excursions, plasma glucose AUC, and plasma glucose AUC excursions after the three main test meals combined | At end of treatment arm or 3 months.
Plasma glucose AUC excursions during a 24 hours when plasma glucose exceeds the following: greater than or equal to 7.5 mmol/L (135 mg/dL), greater than or equal to 7.8 mmol/L (140 mg/dL), and greater than or equal to 10.0 mmol/L (180 mg/dL) | At end of treatment arm or 3 months.
The number of patients with increased plasma glucose during the last 2 hours of each inpatient period | At end of treatment arm or 3 months.
The mean amplitude of glycemic excursion | At end of treatment arm or 3 months.
Concentration of plasma triglycerides and free fatty acids | At end of treatment arm or 3 months.
Self blood glucose monitoring parameters: fasting, premeal, 2 hour postprandial, 2 hour postprandial excursion, bedtime, and overall daily blood glucose value | At end of treatment arm or 3 months.
Insulin dose and body weight | At end of treatment arm or 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Result] Roach P, Malone JK. Comparison of insulin lispro mixture 25/75 with insulin glargine during a 24-h standardized test-meal period in patients with Type 2 diabetes. Diabet Med. 2006 Jul;23(7):743-9. doi: 10.1111/j.1464-5491.2006.01895.x. PMID 16842478
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com